CLINICAL TRIAL: NCT05214261
Title: Laparoscopic-Guided Transversus Abdominis Plane Block Versus Epidural Analgesia in a Colorectal Laparoscopic Surgery. A Protocol for a Randomized Clinical Trial
Brief Title: Laparoscopic-guided TAP Block vs Epidural Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Heikki Huhta, Gastointestinal Surgeon, Adjunct Professor, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112/2021
Record Dates: First submitted 2021-11-16; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Safety; Analgesia, Epidural

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP block group (Experimental): Patiens undergo laparoscopic-guided TAP block installation for laparoscopic clolorectal surgery
  Interventions: Other: Safety and efficiency of post operative analgesia between laparoscopic-assisted TAP block and epidural analgesia
- Epidural analgesia group (Active Comparator): Patients undergo epidural catheters placement for laparoscopic colorectal surgery
  Interventions: Other: Safety and efficiency of post operative analgesia between laparoscopic-assisted TAP block and epidural analgesia

INTERVENTIONS:
Other: Safety and efficiency of post operative analgesia between laparoscopic-assisted TAP block and epidural analgesia — Patients in the TAP group will be given a laparoscopic-assisted TAP block with a total of 2mg/kg of 0.25% bupivacaine in the bilateral subcostal region into four spots of the bilateral subcostal region, two on both sides of the lateral abdomen between the anterior iliac spine and lower costal arch. The TAP block is performed after the first trocar placement before the insertion of other trocars and the beginning of the surgical intervention.
  In the control group epidural catheters will be placed using landmark- and loss-of-resistance techniques while the patient is on the operating table. Infusions of 4ml/h containing 0.125% levobupivacaine and 5.5 μg/mL fentanyl will be started with a CADD Solis VIP-infusion pump at the time of anesthesia induction.

SUMMARY:
The LAPTAP trial will provide evidence on preferred post-operative analgesia method in elective laparoscopic colon surgery.

DETAILED DESCRIPTION:
In most previous studies TAP-block has been inserted by anesthesiologist under ultrasound guidance. TAP blockade can alternatively be performed by a surgeon with laparoscopic visual guidance during trocar placement by aiming injection into fascial plane between the internal oblique and transversus abdominis in the midaxillary line and repeated on the contralateral side. There is lack in studies comparing laparoscopic guided TAP-blockade versus epidural pain analgesia in elective laparoscopic colon surgery exist.

ELIGIBILITY:
IInclusion criteria

* Patients who undergo elective laparoscopic colorectal surgery for colorectal neoplasia, diverticulitis, and other diseases of the colon and rectosigmal area
* Patients able to provide informed written consent
* Patients capable of completing questionnaires at the time of consent

Exclusion criteria

* Documented allergic reaction to morphine, hydromorphone, lidocaine, bupivacaine, fentanyl and/or oxycodone
* Contra-indication to placement of epidural catheter (spinal stenosis, spinal fusion, elevated international normal ratio (INR), anticoagulation, patient refusal, etc.) or TAP block (patient refusal)
* Urgent or emergent surgery precluding epidural catheter placement or TAP block
* Systemic Infection contraindicating epidural catheter placement or TAP block
* Rectal surgery
* Pregnant or suspected pregnancy
* Age < 18 years
* Planned open surgery
* Planned bowel stoma (protective diversion and/or permanent stoma)
* Unwillingness to participate in follow-up assessments
* Patients with severe chronic pain
* Known sensibility for opioid side effects
* i.v.-PCA is contraindicated (for example drug abuse)
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of post-operative hospital stay after elective laparoscopic colorectal surgery. | Up to 1 month
  The primary endpoint in this study is the length of post-operative hospital stay after elective laparoscopic colorectal surgery

SECONDARY OUTCOMES:
Overall operating theatre time | Up to 10 hours
  Overall operating theatre time
Post-operative morphine milligram equivalents recruitments | Up to 1 month
  Post-operative morphine recruiments
Visual analogue scale | Up to 1 month
  The scores range 1 to 10. Higher scores indicates worse outcome in the treatment of anelgesia.
Overall benefit of analgesia score (OBAS) | Up to 1 month
  The scores range 0 - 24. Low OBAS socre indicates high benefit of analgesia
Hospital readmission | 30 and 90-day
  Post-operative readmissions
Time to first flatus | Up to 1 month
  Post-operative flatus
Time to first bowel movement | Up to 1 month
  Post-operative bowel movement
Time to post-operative mobilization | Up to 1 month
  Post-operative mobilization
Overall cost-effectiveness | Up to 6 months
  Overall cost-effectiveness
Post-operative complications related to interventions according to Clavien-Dindo classification | 30 and 90-day
  Post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Huhta, PhD, Principal Investigator — Oulu University Hospital
Locations (1):
- Surgery and Intensive Care Research Unit, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No